CLINICAL TRIAL: NCT00423761
Title: An Open-Label, Single-Sequence Study to Evaluate the Potential CYP 3A4 Pharmacokinetic Interaction of GW876008 in Healthy Subjects
Brief Title: An Investigation To Determine The Potential Interaction Effect Between GW876008 And Midazolam.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRH103152
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics,; tolerability,; healthy,; subjects
MeSH Terms: interventions — Midazolam; GW 876008

INTERVENTIONS:
Drug: midazolam
Drug: GW876008
  Other Names: midazolam

SUMMARY:
This study will evaluate any effect of single and repeated administration of GW876008 on the metabolism of midazolam in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females.
* Normal ECG.
* Agree to remain in the clinic for the time defined in the protocol.
* Subjects must agree to abstain from alcohol for 24 hours prior to the start of dosing until collection of the final pharmacokinetic sample.

Exclusion Criteria:

* Any serious medical disorder or condition.
* Any history of an endocrine disorder.
* Any clinically significant laboratory abnormality.
* History of psychiatric illness.
* Any history of suicidal attempts or behavior.
* Active peptic ulcer disease.
* Positive faecal occult blood.
* The subject smokes or has smoked or has used any nicotine-containing products in the last six months.
* Women having a positive serum HCG pregnancy test at screening, a positive urine pregnancy test before admission to the Unit during the in-house periods, who are not willing to use acceptable methods of contraception or who are lactating or planning to become pregnant within the three months following the screening visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12

PRIMARY OUTCOMES:
Blood levels of GW876008 and midazolam collected on Day 1 of Session 1 and on Days 1 and 14 of Session 2. | on Day 1 of Session 1 and on Days 1 and 14 of Session 2.

SECONDARY OUTCOMES:
12-lead ECG, Continuous Lead II Telemetry & adverse events: day 1 session 1; days 1 & 14 session 2 | day 1 session 1; days 1 & 14 session 2
vital signs & clinical laboratory data: day 1 session 1; days 1, 7 & 14 session 2 | day 1 session 1; days 1, 7 & 14 session 2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MBChB, MFPM, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dallas, Texas, United States